CLINICAL TRIAL: NCT06328374
Title: Prevalence and Detection of Voice and Swallowing Disorders in Adults With and Without Alzheimer's Disease
Brief Title: Voice and Swallowing Disorders in Adults With and Without Alzheimer's Disease
Status: Withdrawn | Type: Observational
Why Stopped: Change of scope of the work given feedback from funding agency leading to new IRB/clinicaltrials.gov registration.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cara Donohue, Ph.D. CCC-SLP, Assistant Professor, Director of Medical Speech-Language Pathology, Vanderbilt University Medical Center
Other Study IDs: 240420
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease; Caregiver Burden; Healthy Aging; Dysphonia; Dysphagia
MeSH Terms: conditions — Alzheimer Disease; Caregiver Burden; Dysphonia; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy community dwelling adults: Healthy adults between the ages of 60-100 with no prior history of neurological, respiratory, or gastrointestinal diseases or swallowing or voice impairments, or history of head and neck surgery, cancer, or radiation to the head or neck will be enrolled in this study.
- Adults with Alzheimer's Disease and their caregivers: Adults with a diagnosis of Alzheimer's disease and their caregivers will be enrolled in this study.

SUMMARY:
This research study is investigating whether people with Alzheimer's disease experience more changes to voice and swallowing than their healthy age-matched peers. The prevalence of swallowing impairments in moderate-severe Alzheimer's Disease is high (85-93%) and voice is also often negatively impacted by Alzheimer's disease. The overall objective of this study is to evaluate the voice and swallowing function of adults with and without Alzheimer's disease. The investigators will also be involving the primary caregivers of individuals with Alzheimer's that are enrolled in the study to better understand the impact of voice and swallowing impairments on the primary caregivers of those with Alzheimer's Disease.

Healthy adults and individuals with Alzheimer's disease will:

* undergo tests of cough, voice, and swallow function
* undergo tests of grip and tongue strength
* complete questionnaires

Caregivers of individuals with Alzheimer's disease will also complete questionnaires.

DETAILED DESCRIPTION:
This study will involve one in-person research visit that will last approximately 1-1.5 hours and will consist of a screening, cough testing, swallow function testing, vocal function testing, assessments of hand grip and tongue strength, and completion of questionnaires. Caregivers of those with Alzheimer's disease will also complete questionnaires at this initial visit.

Following the first research evaluation visit, individuals will be contacted via email or by phone annually for two consecutive years to complete the same questionnaires completed at the initial visit.

ELIGIBILITY:
Healthy Adult Cohort

Inclusion Criteria

1. healthy community dwelling adult (60-100 years old)
2. no prior history of neurological diseases
3. no prior history of respiratory diseases
4. no prior history of head and neck surgery/head and neck cancer/radiation to head and neck region
5. no prior history of swallowing difficulties
6. no prior history of gastroesophageal diseases/impairments
7. absence of vocal fold lesions or paresis/paralysis
8. no recent intubation (≥3 weeks)
9. score ≥26 on the Montreal Cognitive Assessment (MOCA) or the telephone version of the MOCA (t-MOCA)

Exclusion Criteria

1. individual <60 years old, >100 years old
2. history of neurological disease
3. history of respiratory disease
4. history of head and neck surgery/head and neck cancer/radiation to head and neck region
5. history of swallowing difficulties
6. history of gastroesophageal diseases/impairments
7. presence of vocal fold lesions or paresis/paralysis
8. recent intubation (<3 weeks)
9. score <26 on the Montreal Cognitive Assessment (MOCA) or the telephone version of the MOCA (t-MOCA)

AD Cohort

Inclusion Criteria

1. between 60-100 years old
2. diagnosis of AD by neurologist
3. consuming some form of oral intake
4. able to follow basic directions

Exclusion Criteria

1. individual <60 years old, >100 years old
2. diagnosis of another type of dementia
3. not consuming any oral intake
4. unable to follow basic directions

Caregivers of Individuals with AD Cohort

Inclusion Criteria

1. primary caregiver of an individual with AD
2. willing to complete questionnaires/semi-structured interview

Exclusion Criteria

1. not the primary caregiver of an individual with AD
2. unwilling to complete questionnaires/semi-structured interview

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The overall objective of this proposal is to evaluate voice and swallow function in 40 healthy adults and 40 individuals with AD and to evaluate caregiver perceptions of voice and swallow function and burden in 40 caregivers of individuals with AD. Thus, this study will enroll healthy adults, individuals with AD, and caregivers of individuals with AD.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Swallowing safety | During baseline visit at time of enrollment.
  The penetration aspiration scale is a validated 8-point ordinal rating scale that measures the depth of airway invasion and the patient's response during swallowing. Scores range from 1 to 8 with a score of 1 indicating a safe swallow (best score) and 8 indicating silent aspiration (worst score).
Voluntary cough peak expiratory flow | During baseline visit at time of enrollment.
  A measure of cough strength
Vocal fold bowing index | During baseline visit at time of enrollment.
  Vocal fold bowing will be completed as described by Bloch and Behrman.

SECONDARY OUTCOMES:
Swallowing and Eating Related Fatigue Questionnaire (SERF) | During baseline visit at time of enrollment, 1 year after baseline visit, 2 years after baseline visit.
  Scores on the SERF range 0-48 with higher scores indicating greater impairment.
Swallowing Related Quality of Life Questionnaire (SWAL-QOL) | During baseline visit at time of enrollment, 1 year after baseline visit, 2 years after baseline visit.
  Scores on the SWAL-QOL range from 0-100 with lower scores indicating greater impairment.
Voice Handicap Index (VHI) | During baseline visit at time of enrollment, 1 year after baseline visit, 2 years after baseline visit.
  The VHI contains 30 questions, and scores range from 0-120, with higher scores indicating greater perceived voice handicap.
Aging Voice Index (AVI) | During baseline visit at time of enrollment, 1 year after baseline visit, 2 years after baseline visit.
  he AVI consists of 23 questions, with scores ranging from 0-92. Higher scores indicate a greater effect of dysphonia on quality of life.
Grip Strength | During baseline visit at time of enrollment.
  Grip strength be used to quantify clinical frailty using a digital hand dynamometer.
Tongue strength | During baseline visit at time of enrollment.
  Tongue strength will be assessed using the Iowa Oral Pressure Instrument (IOPI).
Clinical frailty scale | During baseline visit at time of enrollment, 1 year after baseline visit, 2 years after baseline visit.
  The clinical frailty scale (scores 1-9) will be used to classify frailty with higher scores indicating greater impairment.
Caregiver Analysis of Reported Experiences with Swallowing Disorders (CARES) Questionnaire | During baseline visit at time of enrollment, 1 year after baseline visit, 2 years after baseline visit.
  Scores on the CARES range from 0-26 with higher scores indicating greater caregiver burden.
Caregiver Self-Assessment Questionnaire | During baseline visit at time of enrollment, 1 year after baseline visit, 2 years after baseline visit.
  Scores range from 0-16 with higher scores indicating greater caregiver burden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT06328374/ICF_001.pdf